CLINICAL TRIAL: NCT03110198
Title: A Randomized, Double-blind Study Investigating the Efficacy and Safety of Mesalazine With Hydrocortisone Sodium Succinate (100mg QD) Enema for 4-Week Treatment in Patients With Ulcerative Colitis (UC)
Brief Title: Mesalazine With Hydrocortisone Sodium Succinate Enema for 4-Week Treatment in Patients With Ulcerative Colitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other); First Affiliated Hospital of Zhongshan Medical University (Other)
Responsible Party: Principal Investigator, Jie Liang, Associated professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20162063-1
Record Dates: First submitted 2017-02-19; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Ulcerative Colitis, Unspecified
Keywords: Mesalazine; Ulcerative Colitis(UC); Enema
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mesalazine with hydrocortisone sodium succinate (Experimental): Mesalazine（4g） with hydrocortisone sodium succinate (100mg ) enema
  Interventions: Drug: Mesalazine with hydrocortisone sodium succinate
- Mesalazine (Active Comparator): Mesalazine （4g）enema
  Interventions: Drug: Mesalazine
- Hydrocortisone sodium succinate (Active Comparator): Hydrocortisone sodium succinate (100mg ) enema
  Interventions: Drug: hydrocortisone sodium succinate

INTERVENTIONS:
Drug: Mesalazine — Mesalazine enema rectal administration at bedtime 4g/100 ml, once daily
  Arms: Mesalazine
Drug: hydrocortisone sodium succinate — hydrocortisone sodium succinate rectal administration at bedtime 100mg/100 ml, once daily
  Arms: Hydrocortisone sodium succinate
Drug: Mesalazine with hydrocortisone sodium succinate — Mesalazine with hydrocortisone sodium succinate rectal administration at bedtime 4g，100mg/100 ml, once daily for induction of remission
  Arms: Mesalazine with hydrocortisone sodium succinate

SUMMARY:
The research aims to evaluate the efficacy and safety of that mesalazine with hydrocortisone sodium succinate for the induction of clinical remission during a 4-week double-blind treatment period in active UC (define as total Mayo score of greater than or equal to 4 and less than or equal to 10). A total of 528 patients will be randomly divided into three group, one will receive mesalazine 4g with hydrocortisone sodium succinate 100mg enema, and the other two group will respectively to receive mesalazine 4g and hydrocortisone sodium 100mg one times daily for 4 weeks. The end of the study for every patient is the improvement of main symptoms.The primary endpoint is the clinical remission after 2 and 4 weeks double-blind treatment, defined on the basis of a total Mayo score ≤ 2 points, with no subscore > 1 point. The secondary endpoint are endoscopic mucosal healing at week 2 and 4 of double-blind period, defined as an absolute subscore for endoscopy portion of the Mayo score of 0 point and the change from baseline in Quality of Life at week 4 of double-blind period based on the IBDQ.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Chinese patients aged ≥18 to ≤ 70 years
2. Newly diagnosed or recurrent active ulcerative colitis (A gold standard for the diagnosis of ulcerative colitis is not available. The diagnosis should be established by a combination of medical history, clinical evaluation, and typical endoscopic and histological findings. An infective cause should be excluded. Where there is doubt about the diagnosis, endoscopic and histological confirmation is necessary after an interval.)
3. Extent of colonic involvement and endoscopy subscore of Mayo score as confirmed by colonoscopy (it should be done within 15 days prior to randomization)
4. Total Mayo score of at least 4 and a score of ≥ 2 for colonoscopy
5. Oralthe stability dose of 5-ASA medicine 14days.
6. Negative stool test at screening to rule out parasites and bacterial pathogens
7. The patient is compliant with Patient Daily Diary
8. Women with childbearing potential must have an efficacious contraception as judged by the investigators and must have a negative pregnancy test result at screening
9. Signed Informed Consent obtained before any trial-related procedures.

Exclusion Criteria:

1. Severe/fulminant ulcerative colitis or toxic dilatation of the colon
2. Prior bowel resection surgery
3. Known infection of human immunodeficiency virus (HIV), Hepatitis B virus (HBV) or Hepatitis C virus (HCV) (Note active Hepatitis B patients should be excluded from the study e.g. HBeAg positive or HBV DNA positive, with the exception for inactive HBsAg carrier)
4. Take the following treatment:

   1. Any 5-ASA enema or suppository therapy during the 14 days prior to screening
   2. Corticosteroids (oral, intravenous, intramuscular, or rectal ) within 7 days prior to screening
   3. Any immunomodulating/suppressive agents during the 60 days prior to screening
   4. Any Anti-TNF therapy during the 6 months prior to screening
   5. Antibiotics (metronidazole and ciprofloxacin) within 7 days prior to screening
   6. Loperamide, nicotine patch and mucilages within 7 days prior to screening
   7. Traditional Chinese Medicine for the treatment of UC (any pharmaceutical form) within 7 days prior to screening
5. Patients allergic to 5-ASA and derivative, any of the excipients, aspirin, or salicylates
6. Known significant hepatic function abnormalities, defined as the values of serum ALT or AST are equal to or more than twice of the upper limit of normal value
7. Women who are planning or actual pregnancy or lactation during study period
8. Alcohol addiction (>40 g of alcohol/day equivalent to >1 L of beer/day, 0.5 L of wine/day, or 6 glasses (2 centiliter, cl) of liquor/day)
9. Drug addiction confirmed by patients' medical history
10. History of disease that would interfere with their participation in the trial, including malignant diseases, bleeding disorders, active gastric or active duodenal ulcers, autoimmune diseases, and mental or emotional disorder
11. Patient participating or having participated in another clinical study 30 days prior to screening
12. Patient who are unlikely to comply with the protocol as judged by the investigator
13. Patients who are unable to fill in the Patient Daily Diary or follow data-capturing procedures
14. Patients with one or more of the diseases: bacillary dysentery, amebic dysentery, chronic schistosomiasis, intestinal tuberculosis and Crohn's disease
15. Patients with any other disease or condition which might interfere with study assessment as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change of clinical remission | 2 weeks, 4 weeks
  Clinical remission after 2 and 4 weeks double-blind treatment, defined on the basis of a total Mayo score ≤ 2 points, with no subscore > 1 point

SECONDARY OUTCOMES:
Change of endoscopic mucosal healing | 2 weeks, 4 weeks
  endoscopic mucosal healing at week 2 and 4 of double-blind period, defined as an absolute subscore for endoscopy portion of the Mayo score of 0 point
Change of quality of life based on the IBDQ | 2 weeks, 4 weeks
  The change from baseline in Quality of Life at week 2 and 4 of double-blind period based on the IBDQ
Change of mental health by Anxiety and Depression Assessment Scale | 2 weeks, 4 weeks
  Assess mental health by Anxiety and Depression Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: jie Liang, professor, Principal Investigator — China,Shaanxi,Xi'an, Xijing Hospital of Digeetive Disease
Locations (1):
- Xijing Digestive Disease, Xi'an, Shaanxi, China